CLINICAL TRIAL: NCT05625464
Title: Effect of Automated Real-time Feedback on Early Sepsis Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Crico (Other)
Responsible Party: Principal Investigator, Kyan Safavi, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020P002676
Record Dates: First submitted 2022-11-13; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Received SCTP monitoring and standard of care
  Interventions: Other: SCTP
- Control (No Intervention): Received standard of care only

INTERVENTIONS:
Other: SCTP — Real-time automated monitoring of the electronic medical record to identify suspected sepsis patients without completion of sepsis bundle measures within 1-hour of the completion deadline and generated reminder pages. Clinicians responsible for patients randomized to the intervention receive reminder pages whereas no pages are sent for control arm patients.
  Arms: Intervention

SUMMARY:
Sepsis is the leading cause of death among US hospitals, accounting for 6% of all hospitalizations and 35% of all inpatient deaths. International guidelines and the CMS SEP-1 bundle stress the importance of adhering to specific steps in the diagnosis and management of sepsis. This can be very difficult, especially in the setting of a busy ED, ward, or ICU where there are multiple simultaneous demands on providers' attention and time. Critical steps can be missed or delayed. The CMS SEP-1 bundle is a measure of compliance with sepsis care that is being tracked nationally across hospitals.

Unfortunately, a recent study demonstrated that every hour of delay to the completion of a sepsis bundle, including antibiotic administration, was associated with a 4% increase in risk-adjusted hospital mortality.

One strategy to improve the care and outcomes of patients with sepsis is the use of information technology to support our providers in a targeted manner. Technology has already been developed and deployed to help with the early identification of patients with sepsis using a Best Practice Alert (BPA), which has been in place at our hospital since 2017. This pop-up window alerts the team to the possibility of sepsis based on data within the medical record. However, once the alert is accepted or declined, the BPA does not offer ongoing support to clinicians, leaving the clinician to track and execute multiple time-based and inter-dependent sepsis bundle measures in a busy, hectic environment. To augment this existing tool, here we propose to study the efficacy of a novel technology called the Sepsis Care Tracking Platform (SCTP) to provide ongoing support at the bedside to providers, thus improving the care we deliver to patients.

SCTP is a monitoring and notification platform that aims to increase the timely delivery of key elements of evidence-based sepsis care. This platform, which was built by clinicians for clinicians, leverages the electronic medical record (EMR) to track real-time compliance with key components of the CMS SEP-1 bundle - timely antibiotics, blood cultures prior to antibiotics, initial lactate, and repeat lactate for those patients with an initially elevated level. SCTP underwent technical validation in Fall 2019 with a pilot in the MGH Emergency Department. The pilot confirmed that SCTP correctly identified missing bundle elements and paged the appropriate team members connected with the patient's care. The pilot also did not find alarm fatigue to be an issue. We hypothesize that SCTP will increase our hospital's compliance with sepsis process metrics and improve patient outcomes.

By monitoring real-time data and automatically alerting bedside providers to missing elements within an actionable timeframe, SCTP has the potential to drive improvements in clinical care even in the extremely busy and complex environment of the emergency department and inpatient units.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 years old and over
2. Who triggered a sepsis best practice advisory that was subsequently acknowledged by a treating clinician as "yes, sepsis possible"

Exclusion Criteria:

1. Transfer from an outside hospital
2. Sepsis best practice advisory triggered while the patient is in an intensive care unit
3. Sepsis best practice advisory triggered while the patient is in a perioperative care area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3269 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
3-hour sepsis bundle order compliance | Within 3 hours of sepsis BPA trigger (time zero)
  Overall 3-hour bundle ordering compliance, defined as orders for all 3-hour bundle measures monitored by the study platform completed within the bundle time limits - i.e., orders for antibiotics, blood cultures, and lactate measurement measured from the electronic medical record at the end of the study period

SECONDARY OUTCOMES:
Antibiotic order compliance | within 3 hours of timezero
  Antibiotic ordering compliance, defined as orders for antibiotics placed within 3 hours of timezero
Blood culture order compliance | within 3 hours of time-zero
  Blood culture ordering compliance, defined as orders for blood cultures placed within 3 hours of time-zero
Initial lactate order compliance | within 3 hours of time-zero
  Initial blood lactate level ordering compliance, defined as orders for initial blood lactate level within 3 hours of time-zero
Repeat lactate order compliance | placed within 6 hours of time-zero and within 3 hours of initial lactate measurement
  Repeat blood lactate level ordering compliance, defined as orders for repeat blood lactate level placed within 6 hours of time-zero and within 3 hours of initial lactate measurement, among patients with initial lactate > 2.0mmol/L
3-hour sepsis bundle care delivery compliance | Within 3 hours of sepsis BPA trigger (time zero)
  Overall 3-hour bundle care delivery compliance, defined as the implementation of all 3-hour bundle measures monitored by the study platform completed within the bundle time limits - i.e., administration of antibiotics, collection of blood cultures prior to antibiotic administration, and lactate measurement.
Antibiotic delivery compliance | within 3 hours of timezero
  Antibiotic delivery compliance, defined as administration of antibiotics within 3 hours of timezero
Blood culture delivery compliance | within 3 hours of timezero and prior to antibiotic administration
  Blood cultures delivery compliance, defined collection of blood cultures within 3 hours of timezero and prior to antibiotic administration
Initial lactate delivery compliance | within 3 hours of time-zero
  Initial lactate delivery compliance, defined measurement of initial lactate within 3 hours of time-zero
Repeat lactate delivery compliance | within 6 hours of time-zero and within 3 hours of initial lactate measurement
  Repeat lactate delivery compliance, defined as the measurement of a repeat lactate within 6 hours of time-zero and within 3 hours of initial lactate measurement, among patients with an initial lactate > 2.0mmol/L
Mortality by Day 28 | Within 28 days of time zero
  Mortality by Day 28
Early mechanical ventilation | within 72 hours of time-zero
  Early mechanical ventilation, defined as the receipt of mechanical ventilation or death within 72 hours of time-zero
Early intensive care unit admission | within 72 hours of time-zero
  Early intensive care unit (ICU) admission, defined as ICU admission or death within 72 hours of time-zero
Mechanical ventilation during hospitalization | within 28 days of time-zero
  Mechanical ventilation during hospitalization, defined as receipt of mechanical ventilation or death within 28 days of time-zero
Early antibiotic discontinuation | at least 24 hours by 48 hours post-time-zero
  Early antibiotic discontinuation, defined as discontinuation of all antibiotics for at least 24 hours by 48 hours post-time-zero
Hospital length of stay | Through day 28 after time zero
  Hospital length of stay, defined as hospital days from time-zero through day 28
Blood culture positivity | 24 hours before or 7 days after time zero
  Blood culture positivity, defined as bacterial growth recovered from any blood culture collected 24 hours before or 7 days after time zero
Non-blood culture positivity | 24 hours before or 7 days after time zero
  Non-blood culture positivity, defined as bacterial pathogen recovery from any urine, respiratory, peritoneal, pleural, joint, or cerebrospinal fluid culture collected 24 hours before or 7 days after time zero
Any culture positivity | 24 hours before or 7 days after time zero
  Any culture positivity, defined as a composite of positive results from either the blood or non-blood culture positivity outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No